CLINICAL TRIAL: NCT01159808
Title: A Study of the Safety and Pharmacokinetics of Single Ascending Oral Doses of INX-08189 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple
Other Study IDs: AI472-001; INH-189-001 (Other: INH-189-001)
Record Dates: First submitted 2010-07-01; First posted 2010-07-09 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Healthy
Keywords: Safety and Pharmacokinetics
MeSH Terms: interventions — BMS-986094

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- INX-08189 (Experimental)
  Interventions: Drug: INX-08189
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INX-08189 — 3, 25 and 100 mg capsules; oral administration, single dose
  Arms: INX-08189
Drug: Placebo — matching placebo capsules, oral administration, single dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the safety of different dose strengths of INX-08189 in healthy adults. The study will also look at how rapidly the drug breaks down in the body (pharmacokinetics or PK). The study objectives include:

* To evaluate the safety of single ascending oral doses of INX-08189 in healthy subjects
* To characterize the pharmacokinetic (PK) profile of single ascending oral doses of INX-08189 in healthy subjects
* To assess the food effect on the PK of a single oral dose of INX-08189

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and post-menopausal (absence of periods for more than 2 years) surgically sterile, or non-pregnant, non-lactating women using a reliable form of contraception (see Inclusion Criteria 9)
2. Age 18 to 65 years, inclusive
3. Normal (no clinically significant abnormalities) laboratory tests (chemistry, hematology and urinalysis)
4. No clinically significant abnormalities on ECG (QTcB interval must be < 450 ms)
5. Weight ≥ 50kg and Body Mass Index (BMI) of 19 to 30, inclusive
6. Negative urine drug screen at screening and on Study Day -1
7. Negative serum βHCG pregnancy test at screening and on Study Day -1 (for all women)
8. Hepatitis B surface antigen, hepatitis C antibody, and HIV antibody negative
9. Agreement to practice a barrier method of birth control plus the use of a spermicide throughout the study period by both male and female subjects (oral contraceptives are not permitted)
10. Able to complete all study visits
11. Signed informed consent form (ICF)

Exclusion Criteria:

1. Any active medical problem for which the subject is being evaluated and/or treated
2. Calculated creatinine clearance (calculated using the IDMS traceable equation for the MDRD value) < 50 mL/min/1.73 m2
3. Regular use of medications, prescription or non-prescription; no medication may be taken within 1 week prior to study dosing
4. Use of alcohol within 48 hours prior to dosing (subjects must also agree to not use alcohol for 96 hours after dosing)
5. Current lactation or breastfeeding
6. Major surgery within 30 days prior to dosing
7. Receipt of an investigational drug within 30 days prior to dosing
8. Donation of blood or plasma within 30 days prior to dosing
9. Any other problem, that in the opinion of the Investigator, will affect the safety of the subject or outcome of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of single ascending oral doses of INX-08189 in healthy subjects | periodically over 14 days
  Safety will be evaluated on the basis of adverse event (AE) incidence, changes in serum chemistry and hematology values, urinalysis results, and changes in vital signs and in electrocardiogram (ECG) findings.
Characterize the pharmacokinetic (PK) profile of single ascending oral doses of INX-08189 in healthy subjects | periodically over 14 days
  Including a determination of maximum observed plasma concentration (Cmax), time at which the maximum plasma concentration was observed (Tmax), time at which concentrations are first measurable in the plasma (Tlag), area under the plasma concentration-time curve from time 0 to time of last measurable plasma concentration (AUC 0-last) and elimination half-life (T 1/2) after single ascending oral doses.
Assess the effect of a high fat meal on the PK parameters | periodically over 14 days
  The effect of food (standard high-fat meal) on the absorption of INX-08189 will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Brian Boehlecke, MD, MSPH, Study Director